CLINICAL TRIAL: NCT03035786
Title: Airway Code Calls - Survey of Management
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Singapore General Hospital (Other)
Collaborators: Tan Tock Seng Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 1607 Airway Code
Record Dates: First submitted 2017-01-24; First posted 2017-01-30 (Estimated); Last update posted 2017-01-30 (Estimated); Status verified 2017-01

CONDITIONS: Intubation; Difficult

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a survey of airway codes, which are emergency mobile phone requests for anaesthetic help to manage acute airway crises in the hospital (out of theatre, out of Surgical Intensive Care Unit, SICU).

The anaesthetists are doctors trained in advance airway management. Patients in the hospital may suffer airway crises e.g. airway obstruction or need for tracheal intubation (insertion of breathing tube) for various reasons. The on call SICU anaesthetists responds to the airway code by attending the patient in need and managing the patient at their own discretion.

Airway management will depend on the anaesthetist's knowledge, skills and experience. it will also depend on the available airway equipment.

We plan to evaluate airway codes for a 24 month period. Parameters include: type of incident; patient factors (including airway assessment); type of equipment used; anaesthetic drugs used; airway management chosen by the attending anaesthetist; and, airway complications.

DETAILED DESCRIPTION:
Airway codes will be managed as standard care. These calls are taken and managed by anaesthetists on call on SICU. The audit form is filled in by the on call anaesthetist after the airway code has been managed. This is an audit looking at:

Primary outcome

•Evaluate the type of airway codes that the SICU anaesthetist is called for

Secondary outcomes:

* Patient factors (including airway assessment)
* Type of equipment used
* Type of anaesthetic drugs used
* Airway management chosen by the attending anaesthetist
* Airway complications.

ELIGIBILITY:
Inclusion Criteria:

* adults outside operating theatre and Surgical Intensive Care Unit requiring emergency anaesthetic airway support

Exclusion Criteria:

* Nil

Ages: 1 Year to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All 'airway code' requests for emergency anaesthetic airway support for adults outside operating theatre and Surgical Intensive Care Unit.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2016-11; Primary Completion 2018-11 (Estimated); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
Survey the type of airway codes that the SICU anaesthetist is called for | One hour post calling of airway code
  Cause of airway codes i.e. respiratory arrest or indication for formal airway management by anaesthetist

SECONDARY OUTCOMES:
Survey of types of equipment needed for airway management | One hour post calling of airway code
  Type of equipment used include airway bag, bougie, videolaryngoscope
Number of participants with predictors of difficult airway | One hour post calling of airway code
  Predictors of difficult airway include small mouth opening, short thyromental distance, prominent upper teeth, receding lower jaw, decreased neck movement, previous surgery, previous radiotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Wong, MBBS FRCA, Principal Investigator — Singapore General Hospital
Locations (2):
- Singapore (2):
  - Singapore General Hospital, Singapore, Singapore
  - Tan Tock Seng Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bowles TM, Freshwater-Turner DA, Janssen DJ, Peden CJ; RTIC Severn Group. Out-of-theatre tracheal intubation: prospective multicentre study of clinical practice and adverse events. Br J Anaesth. 2011 Nov;107(5):687-92. doi: 10.1093/bja/aer251. Epub 2011 Aug 8. PMID 21828342
- [Background] Martin LD, Mhyre JM, Shanks AM, Tremper KK, Kheterpal S. 3,423 emergency tracheal intubations at a university hospital: airway outcomes and complications. Anesthesiology. 2011 Jan;114(1):42-8. doi: 10.1097/ALN.0b013e318201c415. PMID 21150574